CLINICAL TRIAL: NCT05786274
Title: Predicting Cerebrovascular Adverse Events Post Cardiac Surgery With Cardiopulmonary Bypass by Means of Cerebral AutoreguLation Indices
Brief Title: Predicting Cerebrovascular Adverse Events Post Cardiac Surgery
Acronym: PASCAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Vlasta Bari, Principal Investigator, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PASCAL; GR-2021-12372037 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Disease
Keywords: cerebral autoregulation; cardiopulmonary bypass; stroke
MeSH Terms: conditions — Heart Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac surgery with cardiopulmonary bypass patients (Other): Patients will be enrolled before cardiac surgery with cardiopulmonary bypass (CPB) and monitored until after the surgery. Patients enrolled will undergo diffusion weighted magnetic resonance imaging and will be administered with cognitive tests one day before surgery and within one week after surgery. Cerebral blood flow velocity as derived from transcranial Doppler recordings will be acquired from the middle cerebral artery synchronously with arterial pressure, invasively derived from the radial artery, and with the electrocardiogram as derived from patient's monitor. Signals will be acquired before anesthesia induction (BASAL), after anesthesia induction and intubation of the chest (ANESTH) and during CPB (CPB). Each acquisition will last at least 5 minutes and will be prolonged to the maximum possible length in keeping with clinical scheduling. Partial pressure of carbon dioxide and other clinical parameters will be acquired too during the intervention.
  Interventions: Diagnostic Test: Cerebral autoregulation monitoring

INTERVENTIONS:
Diagnostic Test: Cerebral autoregulation monitoring — Perioperative characterization of cerebral autoregulation and autonomic function; characterization of adverse events after surgery

SUMMARY:
The aims of this study are: i) to assess cerebral autoregulation and autonomic control within the different phases of cardiac surgery with cardiopulmonary bypass; ii) to compare cerebral autoregulation measures derived via cerebral blood flow velocity estimated by transcranial Doppler device with simpler measurements derived from near infrared spectroscopy; iii) to develop a predictive model of postoperative cerebrovascular outcome (overt or silent stroke) based on the extracted indices.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* spontaneous sinus rhythm
* no pregnancy
* signed informed consent

Exclusion Criteria:

* age lower than 18 years
* absence of sinus rhythm
* autonomic disorders
* concomitant carotid intervention
* reintervention
* contraindication to MRI
* pregnancy
* impossibility of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Autoregulation index (ARI) | 36 months
  ARI is an index describing the state of cerebral autoregulation from mean cerebral blood velocity and mean arterial pressure. It ranges between 1 and 9. ARI>4 means working autoregulation. ARI<4 means impaired autoregulation. It will be computed for all participants in BASAL, ANESTH, CPB.
Cerebral Oxymetry index (CoX) | 36 months
  CoX is an index describing the state of cerebral autoregulation derived from NIRS and mean arterial pressure. It ranges between 0 and 1. CoX = 1 means perfect coupling. Cox=0 means uncoupling. It will be computed for all participants in BASAL, ANESTH, CPBasurements derived from near infrared spectroscopy
number of patients developing cerebrovascular adverse events | 36 months
  The number of patients developing cerebrovascular adverse events will be assessed by the presence of positive lesions as detected by DW-MRI.

SECONDARY OUTCOMES:
Baroreflex sensitivity | 36 months
  Baroreflex sensitivity will be measured in ms/mmHg. A higher value means a better baroreflex regulation. It will be computed in all participants during BASAL, ANESTH, CPB.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No